CLINICAL TRIAL: NCT03386227
Title: Prophylactic Antibiotics Prior to Embryo Transfer: a Randomized Controlled Trial
Brief Title: Prophylactic Antibiotics Prior to Embryo Transfer (PAPET): RCT
Acronym: PAPET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was prematurely stopped due to extremely low recruitment and lack of feasibility to continue.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: WashingtonU_REI
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Assisted Reproductive Technology; Antibiotic Prophylaxis; Embryo Transfer
Keywords: Assisted Reproductive Technology; Antibiotic Prophylaxis; Microbiome

STUDY DESIGN:
Intervention Model Description: This study will have patients randomized in a 1:1 fashion to antibiotic prophylaxis or withholding antibiotic prophylaxis.
Who Masked: Outcomes Assessor
Masking Description: The embryologists who assess embryo outcomes (as noted in the secondary outcomes) will be blinded to randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prophylactic antibiotics (No Intervention): Current standard of care in our practice for a fresh in vitro fertilization cycle is to administer one dose of 1 gram oral azithromycin on day one of the IVF cycle start to both the male and female partner. In cases of same-sex couples, only the female undergoing the embryo transfer receives prophylaxis. This will serve as our control arm entitled: prophylactic antibiotics.
- No antibiotic prophylaxis. (Experimental): Couples randomized to the no-antibiotic treatment group will not be prescribed oral antibiotic prophylaxis.
  Interventions: Other: Withholding antibiotic prophylaxis

INTERVENTIONS:
Other: Withholding antibiotic prophylaxis — Our intervention will be a deviation from our current standard of care which is universal antibiotic prophylaxis, even in low risk populations. Our intervention will be withholding antibiotic prophylaxis in low risk populations.
  Arms: No antibiotic prophylaxis.

SUMMARY:
The objective of this study is to determine the impact on clinical pregnancy rate of withholding routine prophylactic antibiotic therapy during IVF. The hypothesis is that withholding antibiotic prophylaxis will be non-inferior to routine administration. To test this hypothesis, the investigators will conduct a randomized controlled non inferiority trial. Additionally an exploratory study will be conducted among the first 30 patients undergoing their first cycle enrolled to evaluate the microbiome across the IVF cycle, in addition to the human virome

DETAILED DESCRIPTION:
Over 200,000 in vitro fertilization (IVF) cycles were initiated in the United States in 2015,1 allowing thousands of infertile couples to start families. Although most of the steps in IVF protocols are based on strong evidence, one, prophylactic antibiotic administration, is commonplace but not proven to produce benefit. This practice began in 1978 as a means to prevent bacterial contamination of the tip of the catheter used to transfer embryos into the uterus.2 Although subsequent studies showed that bacterial contamination of the transfer catheters had a negative impact on IVF cycle outcomes,3,4 a more recent, robust randomized controlled trial powered to detect catheter tip contamination rates noted a decrease in contamination with routine administration of amoxicillin-clavulanate but no difference in clinical pregnancy rate.5 Given the limited evidence for benefit and the true risk for subjecting patients to unnecessary treatments, one must determine whether prophylactic antibiotics actually improve the IVF outcome that matters most to couples: pregnancy.

The objective of this study is to determine the impact on clinical pregnancy rate of withholding routine prophylactic antibiotic therapy during IVF. The investigators hypothesis is that withholding antibiotic prophylaxis will be non-inferior to routine administration.

Additionally the investigators propose to conduct a smaller exploratory study in this population of the first 30 women enrolled (15 in each arm) to assess the vaginal microbiome and human virome as obtained by vaginal swab. Existing studies are limited and conflicting regarding influence of the microbiome on IVF cycle outcomes. This would be the first study to evaluate alterations in the vaginal microbiome across the IVF cycle in response to medications and supraphysiologic hormone levels, and the first to evaluate the human virome in this patient population.8 The investigators would examine differences within and between groups and assess for the potential impact and association clinical outcomes of those patients exposed to prophylactic azithromycin, and those who are not. Optimizing the vaginal microbiome could serve as a potential target for therapy to help increase IVF success rates in the future with the goal of a full term, live birth. Samples for male partners will be evaluated as well.

To test the hypothesis, the investigators will conduct a randomized controlled noninferiority trial and pursue the following specific aims:

Specific Aim 1: Determine the effect of withholding prophylactic antibiotic administration on clinical pregnancy rate (defined as a gestational sac, with fetal pole and cardiac activity, on ultrasound).

The investigators hypothesize that withholding prophylactic antibiotics before embryo transfer will be non-inferior (absolute difference ≤15%) to routine prophylaxis in terms of clinical pregnancy rates.

Specific Aim 2: Evaluate the impact of prophylactic antibiotic administration on miscarriage rate (pregnancy loss per clinical pregnancy) before 20 weeks.

The working hypothesis is that miscarriage rates will be equivalent between the two groups.

Specific Aim 3: Determine the effect of no prophylactic antibiotic administration on embryo development.

The investigators hypothesize that embryo development, as evaluated by fertilization rate (number of two-pronuclei embryos per mature oocyte), blastocyst conversion rate (number of day 5 embryos from two-pronuclei embryos), and blastocyst utilization rate (number of day 5 embryos transferred or frozen per two-pronuclei embryos) will be equivalent between the two groups.

Specific Aim 4: Determine the impact of prophylactic antibiotics or withholding prophylaxis on the vaginal and endometrial microbiome.

The investigators hypothesis is that azithromycin will impact the vaginal microbiome. Additionally, it is expected to see changes across the IVF cycle that may be associated with cycle outcome endpoints.

Specific Aim 5: Evaluate the clinical implications of the human virome on IVF outcomes.

The investigators hypothesize that existence of subclinical eukaryotic viruses will be associated with negative IVF cycle outcomes.

Impact: The investigators expect to define the clinical impact of withholding antibiotic prophylaxis before embryo transfer as measured by markers of a successful IVF cycle. As the hypothesis is that withholding prophylaxis will be non-inferior to routine antibiotic administration, these results are expected have a positive clinical impact by decreasing unnecessary broad-spectrum antibiotic exposure and potentially creating a paradigm shift in IVF protocols.

Approach:

This will be a prospective randomized controlled non-inferiority trial in which 178 couples will receive the standard of care prophylactic antibiotics (control) and 178 will not receive prophylactic antibiotics (experimental). The primary outcome is clinical pregnancy rate. The first 50 women enrolled undergoing their first cycle will also be enrolled in the micro biome and virome pilot study as described above. The expected primary outcome is that withholding prophylactic antibiotics will be non-inferior to antibiotic prophylaxis in terms of clinical pregnancy rate with an acceptable non inferiority margin of 15%. Secondary outcomes include spontaneous miscarriage rate and embryo development as measured by fertilization rate, blastocyst conversion rate, blastocyst utilization rate, and live birth rate.Couples with a female partner aged 18-43 years going through a fresh IVF cycle will be recruited. Couples will be excluded from enrollment if they have any contraindication to antibiotic treatment, are not intending to undergo embryo transfer (fertility preservation patients and oocyte donors), require use of extended antibiotic coverage at time of egg retrieval, are already on antibiotics for any reason (ie: upper respiratory infection etc), have a recent history of pelvic infection, or are planning on limited insemination (inseminating a limited number of the eggs retrieved). Couples will only be included in the study once. The primary outcome is clinical pregnancy rate. Secondary outcomes include spontaneous miscarriage rate and embryo development as measured by fertilization rate, blastocyst conversion rate and blastocyst utilization rate and live birth rate.

Couples going through fresh IVF cycles will be identified and their charts reviewed to assess eligibility for inclusion. Couples who meet inclusion criteria will then be contacted via phone by a trained study coordinator and offered enrollment. Those who express interest will have a time arranged for their consent to be signed for both partners. Couples will be randomized after the receipt of signed consent. Randomization to prophylactic antibiotics or no antibiotics will be performed in a block-randomized fashion per cycle number via computer random number generator in a 1:1 ratio. Couples randomized to the antibiotic group will receive the above stated current regimen the day of gonadotropin start. Couples randomized to the no antibiotic treatment group will not be prescribed oral antibiotic prophylaxis. Couples who agree to participate will have their charts marked indicating participation in the study. The couple's respective nurse will receive a message that will remain part of the electronic medical record regarding patient treatment group allocation so they can prescribe antibiotics appropriately. Embryologists will be blinded to patient treatment group allocation.

The expected outcome is that clinical pregnancy rate will be non-inferior without the use of routine antibiotic prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* The female partner must be aged 18-43 years and going through a fresh IVF cycle

Exclusion Criteria:

* Couples will be excluded from enrollment if they have any contraindication to antibiotic treatment, are not intending to undergo embryo transfer (fertility preservation patients and oocyte donors), require use of extended antibiotic coverage at time of egg retrieval, are already on antibiotics for any reason (e.g., upper respiratory infection), have a recent history of pelvic infection, or are planning on limited insemination (inseminating a limited number of the eggs retrieved) or are using donor sperm.

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2018-01-21 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Our primary outcome measure will be obtained at 5-8 weeks gestational age following embryo transfer
  Defined as a gestational sac, with fetal pole and cardiac activity, on ultrasound

SECONDARY OUTCOMES:
Miscarriage rate | Prior to 20 weeks gestation in a previously established clinical pregnancy
  Pregnancy loss per clinical pregnancy before 20 weeks
Embryo development | Intraoperative (This outcome measure will be assessed from the time of egg retrieval to embryo transfer or embryo cryopreservation)
  As evaluated by fertilization rate (number of two-pronuclei embryos per mature oocyte), blastocyst conversion rate (number of day 5 embryos from two-pronuclei embryos), and blastocyst utilization rate (number of day 5 embryos transferred or frozen per two-pronuclei embryos).
Live birth | delivery
  Number of live births per embryo transfer
Reproductive Tract Microbiome | Approximately 30 days from start of IVF cycle
  Swabs will be obtained across the IVF cycle to evaluate changes in the reproductive tract microbiome
Reproductive Tract Virome | Intraoperative (At the time of embryo transfer)
  Swabs will be obtained at the time of embryo transfer to evaluate the virome

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University Reproductive Endocrinology, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kroon B, Hart RJ, Wong BM, Ford E, Yazdani A. Antibiotics prior to embryo transfer in ART. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD008995. doi: 10.1002/14651858.CD008995.pub2. PMID 22419341
- [Background] Brook N, Khalaf Y, Coomarasamy A, Edgeworth J, Braude P. A randomized controlled trial of prophylactic antibiotics (co-amoxiclav) prior to embryo transfer. Hum Reprod. 2006 Nov;21(11):2911-5. doi: 10.1093/humrep/del263. Epub 2006 Jul 10. PMID 16832124
- [Background] Kaye L, Bartels C, Bartolucci A, Engmann L, Nulsen J, Benadiva C. Old habits die hard: retrospective analysis of outcomes with use of corticosteroids and antibiotics before embryo transfer. Fertil Steril. 2017 Jun;107(6):1336-1340. doi: 10.1016/j.fertnstert.2017.04.003. Epub 2017 May 10. PMID 28501367
- [Background] Practice Committee of the American Society for Reproductive Medicine. Electronic address: ASRM@asrm.org; Practice Committee of the American Society for Reproductive Medicine. Performing the embryo transfer: a guideline. Fertil Steril. 2017 Apr;107(4):882-896. doi: 10.1016/j.fertnstert.2017.01.025. PMID 28366416
- [Background] Franasiak JM, Scott RT Jr. Reproductive tract microbiome in assisted reproductive technologies. Fertil Steril. 2015 Dec;104(6):1364-71. doi: 10.1016/j.fertnstert.2015.10.012. Epub 2015 Oct 24. PMID 26597628
- [Background] Fox C, Eichelberger K. Maternal microbiome and pregnancy outcomes. Fertil Steril. 2015 Dec;104(6):1358-63. doi: 10.1016/j.fertnstert.2015.09.037. Epub 2015 Oct 19. PMID 26493119
- [Background] Ledger WJ, Blaser MJ. Are we using too many antibiotics during pregnancy? BJOG. 2013 Nov;120(12):1450-2. doi: 10.1111/1471-0528.12371. No abstract available. PMID 24118809
- [Background] Wylie TN, Wylie KM, Herter BN, Storch GA. Enhanced virome sequencing using targeted sequence capture. Genome Res. 2015 Dec;25(12):1910-20. doi: 10.1101/gr.191049.115. Epub 2015 Sep 22. PMID 26395152
- [Derived] Eskew AM, Stout MJ, Bedrick BS, Riley JK, Herter BN, Gula H, Jungheim ES, Wylie KM. Association of vaginal bacterial communities and reproductive outcomes with prophylactic antibiotic exposure in a subfertile population undergoing in vitro fertilization: a prospective exploratory study. F S Sci. 2021 Feb;2(1):71-79. doi: 10.1016/j.xfss.2021.01.002. Epub 2021 Jan 11. PMID 34632426

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT03386227/Prot_SAP_001.pdf
  • Informed Consent Form: Informed Consent Female Subjects (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT03386227/ICF_002.pdf
  • Informed Consent Form: Informed Consent Male Subjects (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT03386227/ICF_003.pdf